CLINICAL TRIAL: NCT01289444
Title: Longitudinal Pediatric Palliative Care: Quality of Life & Spiritual Struggle
Acronym: FACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maureen Lyon (Other)
Collaborators: St. Jude Children's Research Hospital (Other); Johns Hopkins University (Other); University of Miami (Other); Howard University (Other); Broward Health (Other)
Responsible Party: Sponsor-Investigator, Maureen Lyon, Principal Investigator, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1R01NR012711-01 (NIH)
Record Dates: First submitted 2011-01-28; First posted 2011-02-03 (Estimated); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: HIV
Keywords: palliative care; AIDS; adolescents; quality of life; adherence; spiritual; threat appraisal; treatment congruence; treatment preferences; dialysis; hospitalization; communication; family intervention; Family Centered Advance Care Planning; decision making; advance care planning; end of life
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Communication; Death

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Living Control (Active Comparator): Session 1. Developmental History. Goal: To take a non-medical developmental history. The RA-Control will conduct the session in a structured interview format. Administered, with all medical questions removed to prevent any risk of contamination with the experimental condition.
  Session 2. Safety Tips. Goal: To provide safety information using the American Academy of Pediatrics Bright Futures counseling guides. Participants will be asked questions about seat belt use, etc. Safety information will be provided.
  Session 3. Nutrition Tips. Goal: To provide safety information using the American Academy of Pediatrics Bright Futures nutrition/counseling guides. The Administered by the trained RA-Control to prevent contamination with the FACE condition.
  Interventions: Behavioral: Healthy Living Control
- FAmily CEntered (FACE) ACP (Experimental): Three-60 to 90 minute sessions scheduled one week apart: 1) To assess values, spiritual and other beliefs, and life experiences with illness and EOL care & when to initiate advance care planning. 2) To facilitate conversations and shared decision-making between the adolescent and guardian/surrogate about palliative care & prepare the surrogate to be able to fully represent the adolescent's wishes. 3) Which person the teen wants to make health care decisions for him/her; The kind of medical treatment the teen wants; How comfortable the teen wants to be; How the teen wants people to treat him/her; What teen wants loved ones to know; Any spiritual or religious concerns teens may have.
  Interventions: Behavioral: FAmily CEntered (FACE) ACP

INTERVENTIONS:
Behavioral: FAmily CEntered (FACE) ACP — Three-60 to 90 minute sessions scheduled one week apart: 1) To assess values, spiritual and other beliefs, and life experiences with illness and EOL care & when to initiate advance care planning. 2) To facilitate conversations and shared decision-making between the adolescent and guardian/surrogate about palliative care & prepare the surrogate to be able to fully represent the adolescent's wishes. 3) Which person the teen wants to make health care decisions for him/her; The kind of medical treatment the teen wants; How comfortable the teen wants to be; How the teen wants people to treat him/her; What teen wants loved ones to know; Any spiritual or religious concerns teens may have.
  Other Names: FACE
  Arms: FAmily CEntered (FACE) ACP
Behavioral: Healthy Living Control — Active Comparator: Three 60 to 90 minute sessions scheduled one week apart. 1. Developmental History. Goal: To take a non-medical developmental history. The RA-Control will conduct the session in a structured interview format. Administered with all medical questions removed to prevent any risk of contamination with the experimental condition. 2. Safety Tips. Goal: To provide safety information using the American Academy of Pediatrics Bright Futures counseling guides. Participants will be asked questions about seat belt use, etc. Safety information will be provided.
  3. Nutrition Tips. Goal: To provide safety information using the American Academy of Pediatrics Bright Futures nutrition/counseling guides.
  Other Names: HLC
  Arms: Healthy Living Control

SUMMARY:
Our goal is to advance palliative care to adolescents and their families. We hope our study will decrease suffering (psychological, spiritual, physical) and increase quality of life (QOL). Left unprepared for end-of-life decisions, miscommunication and disagreements may result in families being charged with neglect or court battles over treatment choices. FAmily CEntered (FACE) Advance Care Planning helps prepare adolescents with HIV/AIDS and their families for future medical decisions. We hope to increase families' understanding of their teens' wishes for end-of-life care and to decrease conflict. We will also study communication and spiritual struggle Families will be randomized into the either the Control (N=65 families) or FACE Intervention (N=65 families). FACE families will meet with a trained/certified researcher for three 60- to 90-minute sessions scheduled one week apart: Session 1: Lyon Advance Care Planning Survey© - Adolescent and Surrogate Versions: Session 2: The Respecting Choices Interview® Session 3: Completion of The Five Wishes©. Control families will also meet with a researcher for three 60-to 90-minute sessions scheduled one week apart: Session 1: Developmental History, Session 2: Safety Tips, and Session 3: Nutrition. Questionnaires will be administered five times, when first seen, at 3, 6, 12 and 18 months from the time of Session 3. Hypothesis 1: Compared to an active control, FACE will relieve psychological suffering by 1) increasing congruence in treatment preferences between teens with AIDS and their surrogates, 2) decreasing decisional conflict regarding EOL decision making for future medical treatment in adolescents with AIDS; 3) increasing quality communication about EOL care in adolescent/legal guardian or surrogate dyads; 4) and maximizing QOL.

Hypothesis 2: In addition to the direct effects, FACE will also indirectly affect QOL through dimensions of threat appraisal.

Hypothesis 3: FACE will have stronger effects on the QOL measures among patients who have less spiritual struggle.

Hypothesis 4: Spiritual struggle has both direct and indirect effects on hospitalization/dialysis use. FACE will also affect hospitalization/dialysis use indirectly through threat appraisal and HAART adherence.

DETAILED DESCRIPTION:
Our goal is to advance palliative care with children and their families aimed at relieving suffering (psychological, spiritual, physical) and maximizing quality of life. Left unprepared for end-of-life decisions, miscommunication and disagreements may result in families being charged with neglect, court battles and even legislative intervention. We propose building on our R34, evidence based model, the Family Centered (FACE) Advance Care Planning intervention, to test our full theoretical model examining the putative mediators and moderators, and spiritual struggle (negative religious coping) with a sicker group and adolescents with AIDS in an adequately powered randomized, clinical, 2-arm, controlled trial. FACE is a culturally sensitive and developmentally appropriate, manualized family intervention based on transactional stress and coping theory, which prepares adolescents with HIV/AIDS and their families for end-of-life decision-making through problem solving. Theoretically, threat appraisal is related to Lazarus' concept of primary appraisal, particularly the way in which an event threatens the child's goals or values. Spiritual struggle (negative religious coping) may be a source of distress, causing disparities in palliative care and outcomes. We will test the efficacy of the FACE intervention for increasing communication and congruence in end-of-life treatment preferences between teens with AIDS and their surrogates, and determine if increased congruence can be maintained over time. We will also examine the impact of the FACE intervention on decisional conflict, quality of communication, and patient quality of life. We will also evaluate hypothesized mediators (threat appraisal, HAART adherence) and moderator (spiritual struggle) of study outcomes, including hospitalizations. We will recruit from hospital-based clinics and randomize 130 adolescent/surrogate dyads (N=260 subjects) to either Control (N=65 dyads) or FACE Intervention (N=65 dyads). Participants with HIV dementia, severe depression, suicidality or homicidality or in foster care will not be allowed to participate. Three 60- to 90-minute sessions will be conducted with a certified interviewer at weekly intervals: FACE: Session 1: Lyon Advance Care Planning Survey© - Adolescent and Surrogate Versions: Session 2: The Respecting Choices Interview® Session 3: Completion of The Five Wishes©. Control will also be administered in a family group format to control for time, attention, and Hawthorn effects: Session 1: Developmental History, Session 2: Safety Tips, and Session 3: Safety Tips. Standardized self-report measures will be administered at baseline, immediate post intervention (3 month), and 6, 12 and 18 month post intervention. Generalized estimating equation (GEE) will assess outcomes.

ELIGIBILITY:
Adolescent Inclusion Criteria:

* Diagnosed ever with HIV;
* All ethnic groups;
* Knows HIV status;
* Speaks English;
* Absence of active homicidality or suicidality;
* Absence of HIV dementia;
* IQ >69;
* Consent from the legal guardian for adolescents aged 14-17;
* Consent from the surrogate for adolescents aged 18-21;
* Assent from adolescent aged 14-17;
* Consent from adolescent aged 18-21;
* Absence of severe depression;
* Not in foster care

Legal Guardian Inclusion Criteria for Legal Guardians of Adolescents Age 14-17:

* Adolescent willingness to discuss problems related to HIV/AIDS with them;
* Age 18 or older;
* Ability to speak English;
* Absence of active homicidality, suicidality, or psychosis;
* Absence of HIV dementia;
* Legal guardian;
* Consent to participate; Consent for his/her adolescent to participate;
* Knows HIV status of adolescent;
* Absence of depression in the severe range;

Surrogate Inclusion Criteria for Adolescents Age 18-21:

* Selected by adolescent aged 18 to 21;
* Age 18 or older;
* Willingness to discuss problems related to HIV and end-of-life;
* Absence of active homicidality, suicidality, or psychosis;
* Absence of HIV dementia;
* Speaks English;
* Consent to participate;
* Knows HIV status of adolescent.
* Absence of severe depression;

Exclusion Criteria:

* adolescent or surrogate does not know HIV diagnosis
* being in foster care
* developmentally delayed
* scoring below the cut off on the HIV Dementia Scale
* scoring above the cut off for depressive symptoms on the Beck Depression Inventory
* homicidal, suicidal or psychotic on screening
* does not speak English

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 216 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
congruence in treatment preferences | Change from baseline in Congruence in Treatment Preferences at 18 months post-intervention compared to control
  Measured by the Statement of Treatment Preferences

SECONDARY OUTCOMES:
QOL | Change from baseline in Quality of Life at 18 months post-intervention compared to control
  Measured by score on Varni's Peds QoL
Utilization of hospitalization | Change from baseline in hospitalizations at 18 month follow-up post intervention compared to control
  Hospitalization will be measured by chart review. Each site has hospital based services for patient population
Utilization of dialysis | Change from baseline in use of dialysis at 18 month post-intervention compared to control
  Use of dialysis will be measured by chart review.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen E Lyon, PhD, Principal Investigator — Children's National Research Institute
Locations (5):
- United States (5):
  - Howard University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Diagnostic & Treatment Center (Broward Health), Fort Lauderdale, Florida
  - Univeristy of Miami Miller School of Medicine, Miami, Florida
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be shared upon request to the PI after the close of the study.
Supporting Information: Study Protocol, SAP
Time Frame: September 1, 2017 to September 1, 2020
Access Criteria: Graduate students in accredited programs, residents, fellows, faculty in accredited programs.

REFERENCES:
- [Background] Lyon ME, Garvie PA, Briggs L, He J, McCarter R, D'Angelo LJ. Development, feasibility, and acceptability of the Family/Adolescent-Centered (FACE) Advance Care Planning intervention for adolescents with HIV. J Palliat Med. 2009 Apr;12(4):363-72. doi: 10.1089/jpm.2008.0261. PMID 19327074
- [Background] Lyon ME, Garvie PA, McCarter R, Briggs L, He J, D'Angelo LJ. Who will speak for me? Improving end-of-life decision-making for adolescents with HIV and their families. Pediatrics. 2009 Feb;123(2):e199-206. doi: 10.1542/peds.2008-2379. PMID 19171571
- [Background] Lyon ME, Garvie PA, Briggs L, He J, Malow R, D'Angelo LJ, McCarter R. Is it safe? Talking to teens with HIV/AIDS about death and dying: a 3-month evaluation of Family Centered Advance Care (FACE) planning - anxiety, depression, quality of life. HIV AIDS (Auckl). 2010;2:27-37. doi: 10.2147/hiv.s7507. Epub 2010 Feb 18. PMID 22096382
- [Background] Lyon ME, Garvie PA, Briggs L, He J, D'Angelo LJ, McCarter R. (September, 2010 on line, in press). Does spirituality protect psychological adjustment, quality of life or medication adherence when talking to HIV+ Adolescents about death and dying? Journal of Adolescent Health.
- [Background] Wilkins ML, Dallas RH, Fanone KE, Lyon ME. Pediatric palliative care for youth with HIV/AIDS: systematic review of the literature. HIV AIDS (Auckl). 2013 Jul 29;5:165-79. doi: 10.2147/HIV.S44275. Print 2013. PMID 23930080
- [Background] Rosenberg AR, Wolfe J, Wiener L, Lyon M, Feudtner C. Ethics, Emotions, and the Skills of Talking About Progressing Disease With Terminally Ill Adolescents: A Review. JAMA Pediatr. 2016 Dec 1;170(12):1216-1223. doi: 10.1001/jamapediatrics.2016.2142. PMID 27749945
- [Background] Lee BC, et al. Who Will Speak for Me? Disparities in Palliative Care Research with Unbefriended Adolescents Living with HIV/AIDS. Journal of Palliative Medicine. 20(10), 2017. doi: 10.1089/jpm.207.0053
- [Result] Dallas RH, Wilkins ML, Wang J, Garcia A, Lyon ME. Longitudinal Pediatric Palliative Care: Quality of Life & Spiritual Struggle (FACE): design and methods. Contemp Clin Trials. 2012 Sep;33(5):1033-43. doi: 10.1016/j.cct.2012.05.009. Epub 2012 Jun 1. PMID 22664645
- [Result] Dallas RH, Kimmel A, Wilkins ML, Rana S, Garcia A, Cheng YI, Wang J, Lyon ME; Adolescent Palliative Care Consortium.. Acceptability of Family-Centered Advanced Care Planning for Adolescents With HIV. Pediatrics. 2016 Dec;138(6):e20161854. doi: 10.1542/peds.2016-1854. Epub 2016 Nov 1. PMID 27940700
- [Result] Lyon ME, Kimmel AL, Cheng YI, Wang J. The Role of Religiousness/Spirituality in Health-Related Quality of Life Among Adolescents with HIV: A Latent Profile Analysis. J Relig Health. 2016 Oct;55(5):1688-99. doi: 10.1007/s10943-016-0238-3. PMID 27071797
- [Result] Lyon ME, D'Angelo LJ, Dallas RH, Hinds PS, Garvie PA, Wilkins ML, Garcia A, Briggs L, Flynn PM, Rana SR, Cheng YI, Wang J. A randomized clinical trial of adolescents with HIV/AIDS: pediatric advance care planning. AIDS Care. 2017 Oct;29(10):1287-1296. doi: 10.1080/09540121.2017.1308463. Epub 2017 Mar 30. PMID 28359212
- [Result] Lyon ME, Dallas RH, Garvie PA, Wilkins ML, Garcia A, Cheng YI, Wang J; Adolescent Palliative Care Consortium. Paediatric advance care planning survey: a cross-sectional examination of congruence and discordance between adolescents with HIV/AIDS and their families. BMJ Support Palliat Care. 2019 Mar;9(1):e22. doi: 10.1136/bmjspcare-2016-001224. Epub 2017 Sep 21. PMID 28935629
- [Result] Lyon ME, Garvie PA, D'Angelo LJ, Dallas RH, Briggs L, Flynn PM, Garcia A, Cheng YI, Wang J; Adolescent Palliative Care Consortium. Advance Care Planning and HIV Symptoms in Adolescence. Pediatrics. 2018 Nov;142(5):e20173869. doi: 10.1542/peds.2017-3869. Epub 2018 Oct 19. PMID 30341154
- [Result] Lyon ME, D'Angelo LJ, Cheng YI, Dallas RH, Garvie PA, Wang J; Adolescent Palliative Care Consortium. The influence of religious beliefs and practices on health care decision-making among HIV positive adolescents. AIDS Care. 2020 Jul;32(7):896-900. doi: 10.1080/09540121.2019.1668523. Epub 2019 Sep 19. PMID 31535560